CLINICAL TRIAL: NCT04101942
Title: Internet-delivered Prolonged Exposure Provided Soon After Traumic Events: An Efficacy Trial
Brief Title: An Internet-delivered Cognitive-behavioral Intervention Provided Soon After Trauma: a RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, PhD, licensed psychologist, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPN
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based CBT (Experimental): The experimental group will go through active internet-based treatment which is delivered on a safe internet platform. Treatment is divided into four modules, each containing homework assignments. Participants in the experimental group will be assigned a therapist that they can contact through a message system in the platform and expect answer within 36 hours on weekdays
  Interventions: Behavioral: Internet-based CBT
- Control condition (assessment only) (No Intervention): Waitlist control, i.e. no active active intervention during waiting list period. Will be offered treatment after 7 weeks.

INTERVENTIONS:
Behavioral: Internet-based CBT — The experimental group will go through active internet-based treatment which is delivered on a safe internet platform. Treatment is divided into four modules, each containing homework assignments. Participants in experimental group will be assigned a therapist that they can contact through a message system in the platform and expect answer within 36 hours.
  Arms: Internet-based CBT

SUMMARY:
The primary objective with this study is to investigate the short-term efficacy (primary endpoint at week 3) of Internet-delivered cognitive behavior therapy (ICBT) provided soon after trauma. The secondary objective is to investigate the long-term efficacy (primary endpoint at week 7) of ICBT. 100 participants recently exposed to a potentially traumatic event will be randomised to either ICBT or assessment only.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

The primary objective with this study is to investigate the short-term efficacy (primary endpoint at week 3) of Internet-delivered cognitive behavior therapy (ICBT) provided soon after trauma.

SECONDARY OBJECTIVES The secondary objective is to investigate the long-term efficacy (primary endpoint at week 7) of ICBT.

Trial design: Randomized trial where participants are allocated to either ICBT (n=50) or control group (assessment only; n=50). Participants randomized to control group are subsequently offered identical ICBT treatment, so that all participants will eventually receive treatment.

All participants are assessed at baseline (W0), post-treatment (primary endpoint; W3) and at one-month follow-up (secondary endpoint; W7). Long-term follow-up assessments are also conducted at 6- and 12-months. The primary outcome measure is also measured weekly from baseline and up to the 1-month follow-up (W7).

Primary outcome measure used are the Posttraumatic Stress Disorder Checklist for Diagnostic and Statical Manual, Fifth Edition (PCL-5). Secondary outcome measures used are Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S), Euroqol (EQ-5D) and Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P).

Participants are self-referred through advertisements in newspapers, web-pages, social media and at primary care, psychiatric and emergency clinics throughout Sweden. Interested applicants do an Internet-administered screening on an encrypted webpage using the PCL-5, MADRS-S, Alcohol User Disorders Identification Test (AUDIT), Drug User Disorders Identification Test (DUDIT), TIC-P, questions about inclusion and exclusion criteria and also give general background information. Written information about the study is given including objectives, benefits, risks and requirements imposed by the study.

An assessor calls the participant and conducts a structured clinical interview including The Mini-International Neuropsychiatric Interview (M.I.N.I.). The aim of this interview is to preliminary assess inclusion criteria and rule out exclusion criteria. Information is also given over the phone by the interviewer about the study protocol.

Safety parameters Participants will have the opportunity to report any adverse events during treatment, at posttreatment and follow-up assessment.

Data collection: Data will be collected electronically via the treatment platform.

Main statistical analysis: Between-group estimates on outcome are done using a mixed-effects regression model with repeated measurements. All analyses will be done according to intention to treat and post hoc per protocol analyses will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* • Experienced psychological trauma in the past two months according to criterion A for PTSD in the DSM-5 (exposed to death, threatened death, actual or threatened serious injury, or actual or threatened sexual violence).

  * At least mild clinical symptoms assessed using the PCL-5
  * ≥ 18 years
  * Situated in Sweden
  * Informed consent

Exclusion Criteria:

* Other serious comorbidity as primary concern (ongoing substance dependence, untreated bipolar disorder, psychotic symptoms, severe depression, borderline personality disorder, high suicidal risk according to the M.I.N.I.)
* Not fluent speaking in Swedish
* Receiving CBT for trauma-related symptoms
* Ongoing trauma-related threat (e.g. living with a violent spouse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2020-09-06 (Actual)

PRIMARY OUTCOMES:
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Baseline, weekly from baseline up to 1-month follow-up, 6 month follow up and 12 month follow up
  Change in symptoms of post traumatic stress from baseline, during treatment to post treatment and follow up (6 and 12 months). The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. All items are scored on a 0-4 scale. Higher score indicate worse severity.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S) | Baseline, post treatment week 3, one-month follow up, 6 month follow up and 12 month follow up
  Change in depressive symptoms from baseline to post treatment and follow up (1, 6 and 12 months). The Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S) is a 9 item self-report measure that assesses the presence and severity of depressive symptoms. All items are scored on a 0-6 scale. Higher score indicate worse severity.
Euroqol, EQ-5D | Baseline, post treatment week 3, one-month follow up, 6 month follow up and 12 month follow up
  Change in overall health from baseline to post treatment and follow up (1, 6 and 12 months). EQ-5D is a standardised self-report measure of overall health status measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a three-level scale: 1 having no problems, 2 having some problems and 3 having extreme problems. A higher score indicate worse severity.
Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | Baseline, post treatment week 3, one-month follow up, 6 month follow up and 12 month follow up
  Change in economic costs from baseline, post treatment, 1 month, 6 month and 12 months follow up. TIC-P collect data on medical consumption and productivity losses in patients with mild to moderate mental health problems. A higher score indicate worse severity.
Adverse Events | Baseline, post treatment week 3, one-month follow up, 6 month follow up and 12 month follow up
  Number of adverse events from baseline, 1 month, 6 month and 12 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Andersson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No